CLINICAL TRIAL: NCT02798133
Title: Open Lung Approach Versus Standard Protective Strategies: Effects on Driving Pressure and Ventilatory Efficiency During Anesthesia
Brief Title: Open Lung Approach Versus Standard Protective Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Carlos Ferrando, MD, PhD, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OLA
Record Dates: First submitted 2016-06-05; First posted 2016-06-14 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Lung Collapse
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OLA (Experimental): recruitment maneuver + individualized PEEP
  Interventions: Procedure: OLA
- RM-5 (Active Comparator): recruitment maneuver + fixed standard PEEP
  Interventions: Procedure: RM-5

INTERVENTIONS:
Procedure: OLA — PEEP titration trial for best Cdyn after the alveolar recruitment maneuver
  Arms: OLA
Procedure: RM-5 — Fixed standard PEEP after the alveolar recruitment maneuver
  Arms: RM-5

SUMMARY:
The aim of this study was to compare the effects of adding a recruitment maneuver (RM) to low tidal volume (VT) ventilation, with or without an individualized post-RM positive end-expiratory pressure (PEEP) setting in lung-healthy patients during anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III undergoing elective major abdominal surgery including pancreatic-duodenectomy, gastrectomy and liver resection

Exclusion Criteria:

* i) laparoscopic surgery, ii) patients with previous respiratory disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
driving pressure | intraoperative
  The driving pressure is a physiological ventilatory parameter measured as platteau pressure minus PEEP. This parameter may be associated with postoperative pulmonary complications

SECONDARY OUTCOMES:
ventilatory efficiency | intraoperative
  Ventilatory efficiency measured with volumetric capnography which includes dead space and tidal elimination of carbon dioxide.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Neto AS, Hemmes SN, Barbas CS, Beiderlinden M, Fernandez-Bustamante A, Futier E, Gajic O, El-Tahan MR, Ghamdi AA, Gunay E, Jaber S, Kokulu S, Kozian A, Licker M, Lin WQ, Maslow AD, Memtsoudis SG, Reis Miranda D, Moine P, Ng T, Paparella D, Ranieri VM, Scavonetto F, Schilling T, Selmo G, Severgnini P, Sprung J, Sundar S, Talmor D, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Amato MB, Costa EL, de Abreu MG, Pelosi P, Schultz MJ; PROVE Network Investigators. Association between driving pressure and development of postoperative pulmonary complications in patients undergoing mechanical ventilation for general anaesthesia: a meta-analysis of individual patient data. Lancet Respir Med. 2016 Apr;4(4):272-80. doi: 10.1016/S2213-2600(16)00057-6. Epub 2016 Mar 4. PMID 26947624
- [Background] Kacmarek RM, Villar J, Sulemanji D, Montiel R, Ferrando C, Blanco J, Koh Y, Soler JA, Martinez D, Hernandez M, Tucci M, Borges JB, Lubillo S, Santos A, Araujo JB, Amato MB, Suarez-Sipmann F; Open Lung Approach Network. Open Lung Approach for the Acute Respiratory Distress Syndrome: A Pilot, Randomized Controlled Trial. Crit Care Med. 2016 Jan;44(1):32-42. doi: 10.1097/CCM.0000000000001383. PMID 26672923
- [Background] Ferrando C, Mugarra A, Gutierrez A, Carbonell JA, Garcia M, Soro M, Tusman G, Belda FJ. Setting individualized positive end-expiratory pressure level with a positive end-expiratory pressure decrement trial after a recruitment maneuver improves oxygenation and lung mechanics during one-lung ventilation. Anesth Analg. 2014 Mar;118(3):657-65. doi: 10.1213/ANE.0000000000000105. PMID 24557111
- [Derived] Ferrando C, Suarez-Sipmann F, Tusman G, Leon I, Romero E, Gracia E, Mugarra A, Arocas B, Pozo N, Soro M, Belda FJ. Open lung approach versus standard protective strategies: Effects on driving pressure and ventilatory efficiency during anesthesia - A pilot, randomized controlled trial. PLoS One. 2017 May 11;12(5):e0177399. doi: 10.1371/journal.pone.0177399. eCollection 2017. PMID 28493943